CLINICAL TRIAL: NCT00342602
Title: Influence of Host Genetic Factors in Development of PML in an AIDS Cohort
Brief Title: Genetics of Progressive Multifocal Leukoencephalopathy and Acquired Immunodeficiency Syndrome
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Multicenter AIDS Cohort Study (MACS) (Unknown)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905218; 05-C-N218
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2006-06

CONDITIONS: PML; AIDS
Keywords: JC Virus; Opportunistic Infection; Single Nucleotide Polymorphism; Genotype; Sequencing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opportunistic Infections

SUMMARY:
This study will identify genetic factors associated with the development of progressive multifocal leukoencephalopathy (PML) in patients with acquired immunodeficiency syndrome (AIDS). PML is a life-threatening infection of the brain that affects about 5 percent of untreated patients with AIDS. Its symptoms include mental deterioration, vision loss, speech disturbances, ataxia (inability to coordinate movements), paralysis, and coma. PML is caused by a polyomavirus called the JC virus.

It is estimated that up to 80 percent of the human population has been exposed to the JC virus, but the disease is very rare. The virus only becomes active in people who have compromised immune systems, such as those undergoing immune suppressive chemotherapy for cancer and those with damaged immune systems due to HIV.

Patients who have participated in the Multicenter AIDS Cohort Study may be eligible for this study, as well as healthy normal volunteers who will serve as controls. The study will review clinical information from patients and analyze genetic factors from both patients and control subjects to investigate genes associated with AIDS and JC virus infection.

DETAILED DESCRIPTION:
The purpose of this study is to identify host genetic factors that contribute to the development of Progressive Multifocal Leukoencephalopathy (PML) associated with JC virus. JC virus is one of many opportunistic infections that arise in AIDS patients. JC virus is widely distributed in the general population, with estimates of population exposure ranging from 30-80%. JC virus remains latent in the host, and in profoundly immunosuppressed patients, JC virus can cause PML, a fatal disease associated with neurotropic JC virus that lytically infects oligodendrocytes. In untreated AIDS populations, the frequency of PML has been estimated at roughly 5%. This study will identify host genetic factors that may contribute to the development of PML in the AIDS population.

ELIGIBILITY:
* No available subjects will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, Los Angeles, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - Johns Hopskins Hospital, Baltimore, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Berger JR, Kaszovitz B, Post MJ, Dickinson G. Progressive multifocal leukoencephalopathy associated with human immunodeficiency virus infection. A review of the literature with a report of sixteen cases. Ann Intern Med. 1987 Jul;107(1):78-87. doi: 10.7326/0003-4819-107-1-78. PMID 3296901